CLINICAL TRIAL: NCT04895436
Title: A Multicenter, Open-Label, Phase 2 Study to Evaluate the Efficacy and Safety of Venetoclax-Obinutuzumab Retreatment in Patients With Recurring Chronic Lymphocytic Leukemia
Brief Title: Study to Assess Change in Disease Activity and Adverse Events of Oral Venetoclax With Intravenous (IV) Obinutuzumab in Adult Participants With Recurring Chronic Lymphocytic Leukemia (CLL)
Acronym: ReVenG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: F. Hoffmann-La Roche Ltd; German CLL Study Group (GCLLSG); Dana-Farber Cancer Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20-356; 2023-504599-10-00 (Other: EU CT)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2021-05-19; First posted 2021-05-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Chronic Lymphocytic Leukemia (CLL); Venetoclax; ABT-199; Venclexta; GDC-0199; Obinutuzumab; Gazyva; GA101; Cancer; ReVenG
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — venetoclax; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 - venetoclax + obinutuzumab (Experimental): Participants will receive venetoclax + obinutuzumab for six 28-day cycles followed by venetoclax for six 28-day cycles.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab
- Cohort 2 - venetoclax + obinutuzumab (Experimental): Participants will receive venetoclax + obinutuzumab for six 28-day cycles followed by venetoclax for eighteen 28-day cycles.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Venetoclax — Oral tablet
  Other Names: Venclexta; ABT-199; GDC-0199
Drug: Obinutuzumab — Intravenous (IV) infusion
  Other Names: GA101; Gazyva

SUMMARY:
Chronic lymphocytic leukemia (CLL) is the most common leukemia (cancer of blood cells). The purpose of this study is to assess retreatment with venetoclax-obinutuzumab (VenG) in participants previously treated with fixed duration first-line (IL) therapy of venetoclax in combination with an anti-CD20 antibody +/- X (where X is any additional drug). Adverse events and change in disease activity will be assessed.

Venetoclax is an approved drug for the treatment of CLL. Study doctors put the participants in 1 of 2 groups, called cohorts, based on when symptoms of CLL came back after previous treatment in first-line. Approximately 75 adult participants with CLL who have been treated with venetoclax in combination with an anti-CD20 antibody +/- X will be enrolled in the study in approximately 60 sites worldwide.

Participants will receive intravenous (IV) obinutuzumab + oral venetoclax (VenG) in 28-day cycles for a total of 6 cycles per cohort, followed by 6 to 18 cycles of venetoclax alone, for a total treatment of 12 to 24 cycles, depending on the cohort.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of chronic lymphocytic leukemia (CLL) that requires treatment for CLL according to International Workshop for Chronic Lymphocytic Leukemia (iwCLL) 2018 criteria.
* Previously completed venetoclax + anti-CD20 antibody +/- X regimen as a fixed duration first-line (1L) therapy and achieved documented response, defined as complete remission, complete remission with incomplete marrow recovery, partial remission, or nodular partial remission.
* More than 24 months (Cohort 1) or 12-24 months (Cohort 2) have elapsed between last dose of venetoclax and disease progression after completion of 1L treatment.

Exclusion Criteria:

- Received intervening treatment for CLL after completing previous treatment with a venetoclax + anti-CD20 antibody +/- X regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Overall response (OR) in Cohort 1 after end of combination treatment | 9 months
  OR is defined as the percentage of participants achieving a best response of partial remission (PR), nodular partial remission (nPR), complete remission with incomplete marrow recovery (CRi), or complete remission (CR). Disease assessments will be based on the 2018 International Workshop for Chronic Lymphocytic Leukemia (iwCLL) criteria for tumor response.

SECONDARY OUTCOMES:
OR in Cohort 1 after end of combination treatment | 9 months
  OR rate is defined as the percentage of participants achieving a best response of CR or CRi
OR in Cohort 1 after end of treatment | 15 months
  OR is defined as the percentage of participants achieving a best response of PR, nPR, CRi, or CR. Disease assessments will be based on the 2018 iwCLL criteria for tumor response.
Time to Response (TTR) in Cohort 1 | 15 months
  TTR is defined as the time from first dose until first response (PR or better).
Duration of Response (DOR) in Cohort 1 | 15 months
  DOR is defined as the time from first response (PR or better) until progressive disease (PD) or death.
Time to Next Treatment (TTNT) for CLL in Cohort 1 | 15 months
  TTNT is defined as the time from first dose until first dose of a non-protocol anti-CLL therapy.
Progression-free Survival (PFS) in Cohort 1 | 15 months
  PFS is defined as the time from first dose until PD or death.
Overall Survival (OS) in Cohort 1 | 15 months
  OS is defined as the time from first dose until death.
Percentage of Participants with Undetectable Minimal Residual Disease (uMRD) rate (<10^-4) in Cohort 1 after end of combination treatment | 9 months
  Percentage of participants with uMRD rate, measured in peripheral blood.
Percentage of Participants with Undetectable Minimal Residual Disease (uMRD) rate (<10^-4) in Cohort 1 after end of treatment | 15 months
  Percentage of participants with uMRD rate, measured in peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (58):
- United States (15):
  - Moores Cancer Center at UC San Diego /ID# 230157, La Jolla, California
  - Winship Cancer Institute of Emory University /ID# 230643, Atlanta, Georgia
  - Des Moines Oncology Research Association /ID# 232606, Des Moines, Iowa
  - Dana-Farber Cancer Institute /ID# 230061, Boston, Massachusetts
  - Henry Ford Hospital /ID# 230268, Detroit, Michigan
  - St. Lukes Hospital of Duluth /ID# 250021, Duluth, Minnesota
  - Hattiesburg Clinic /ID# 233443, Hattiesburg, Mississippi
  - Summit Medical Group-Florham Park /ID# 244782, Florham Park, New Jersey
  - Regional Cancer Care Associates /ID# 244620, Hackensack, New Jersey
  - University of North Carolina /ID# 233313, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center /ID# 230201, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center /ID# 249533, Winston-Salem, North Carolina
  - The Ohio State University /ID# 230439, Columbus, Ohio
  - Pennsylvania Oncology Hematolo /ID# 249637, Philadelphia, Pennsylvania
  - University of Wisconsin-Madiso /ID# 232612, Madison, Wisconsin
- Australia (3):
  - Royal Adelaide Hospital /ID# 229898, Adelaide, South Australia
  - Northern Hospital Epping /ID# 229847, Epping, Victoria
  - Peter MacCallum Cancer Ctr /ID# 254634, Melbourne, Victoria
- Austria (7):
  - Universitaetsklinikum St. Poelten /ID# 243493, Sankt Pölten, Lower Austria
  - Landeskrankenhaus Hochsteiermark, Standort Leoben /ID# 267569, Leoben, Styria
  - Ordensklinikum Linz GmbH Barmherzige Schwestern /ID# 249516, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 230013, Vienna, Vienna
  - Klinik Ottakring /ID# 230019, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 230015, Salzburg
  - Hanusch Krankenhaus /ID# 230010, Vienna
- Brazil (3):
  - Hospital de Clinicas de Porto Alegre /ID# 243657, Porto Alegre, Rio Grande do Sul
  - Hospital Nove de Julho /ID# 243658, São Paulo, São Paulo
  - Instituto de Ensino e Pesquisas Sao Lucas /ID# 243659, São Paulo
- Bulgaria (2):
  - UMHAT Sveti Georgi EAD /ID# 272321, Plovdiv
  - MHAT Hristo Botev /ID# 229687, Vratsa
- Germany (17):
  - Stauferklinikum Schwaebisch Gmuend /ID# 230176, Mutlangen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 230164, Ulm, Baden-Wurttemberg
  - VK&K Studien GbR /ID# 230198, Landshut, Bavaria
  - Muenchen Klinik Schwabing /ID# 230197, Munich, Bavaria
  - Universitaetsmedizin Rostock /ID# 230190, Rostock, Mecklenburg-Vorpommern
  - Universitaetsklinikum Koeln /ID# 230296, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum des Saarlandes /ID# 248747, Homburg, Saarland
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf /ID# 230168, Dresden, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 230186, Kiel, Schleswig-Holstein
  - Onkologische Schwerpunktpraxis /ID# 245465, Berlin
  - Charite Universitaetsmedizin Berlin Campus Virchow-Klinikum /ID# 248748, Berlin
  - Duplicate_DIAKO Ev. Diakonie-Krankenhaus gemeinnuetzige GmbH /ID# 230238, Bremen
  - Universitaetsklinikum Essen /ID# 230181, Essen
  - Universitaetsklinikum Halle (Saale) /ID# 245350, Halle
  - OncoResearch Lerchenfeld GmbH /ID# 230191, Hamburg
  - Klinikum Landshut AdöR der Stadt Landshut /ID# 242991, Landshut
  - Bruederkrankenhaus St. Josef Paderborn /ID# 230177, Paderborn
- Israel (4):
  - Hadassah /ID# 245059, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 243219, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 243218, Tel Aviv, Tel Aviv
  - Rabin Medical Center. /ID# 243220, Petah Tikva
- Italy (2):
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 229504, Turin, Piedmont
  - Azienda Ospedaliera Santa Maria Terni /ID# 229442, Terni
- Fundeni Clinical Institute /ID# 241614, Bucharest, București, Romania
- Hospital Universitario de la Princesa /ID# 229665, Madrid, Spain
- United Kingdom (3):
  - Blackpool Victoria Hospital /ID# 267280, Blackpool, Lancashire
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 250733, Norwich, Norfolk
  - Leeds Teaching Hospitals NHS Trust /ID# 250732, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/